CLINICAL TRIAL: NCT02997137
Title: Impact of a Specific Amino Acid Composition With Micronutrients on Wellbeing and Endocrine-cardiometabolic Situation of Patients With Chronic Exhaustion Conditions, Such as Burnout
Brief Title: Impact of an Amino Acid Composition With Micronutrients on Wellbeing of Patients With Chronic Exhaustion Conditions
Acronym: BOT-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Doris Meister (Industry)
Responsible Party: Sponsor-Investigator, Doris Meister, Doris Meister, Sponsor-Investigator, Kyberg Vital GmbH
Organization: Kyberg Vital GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Kyberg-03
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Psychological Distress
Keywords: Chronic psychological distress; Chronic exhaustion conditions; Perceived Stress Questionnaire 30 (PSQ30); Stress management; Dietary supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOT-01 (Active Comparator): Dietary supplement: specific amino acid composition with micronutrients
  Interventions: Dietary Supplement: BOT-01
- Placebo (Placebo Comparator): Placebo contains no amino acids and no micronutrients and is identical in appearance and solution properties
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: BOT-01 — Amino acid composition with micronutrients, once a day (in the morning) content of a sachet mixed with 200 ml water.
  Duration: 12 weeks
  Other Names: Brand name: aminoplus burnout
  Arms: BOT-01
Other: Placebo — Placebo, once a day (in the morning) content of a sachet mixed with 200 ml water.
  Placebo contains no amino acids and micronutrients and is identical in appearance and solution properties.
  Duration: 12 weeks
  Arms: Placebo

SUMMARY:
Chronic psychological distress can lead to chronic exhaustion conditions, such as burnout. These conditions are associated with a deficiency of specific amino acids and micronutrients that cause endocrine-cardiometabolic abnormalities. These people have specific medically-determined nutrient requirements.

Aim of this study is to demonstrate, that the daily oral administration of a specific amino acid composition (dosage 4.2 g/day) with micronutrients (e. g. 7 vitamins of the B-complex, magnesium, zinc) designed to decrease chronic exhaustion conditions will significantly decrease the perceived chronic distress and associated chronic exhaustion conditions of women and men after 8 and 12 weeks.

DETAILED DESCRIPTION:
Chronic psychological distress can lead to chronic exhaustion conditions, such as burnout. This clinical condition is characterized by reduced satisfaction in performance, exhaustion and depersonalization. Individuals under prolonged exposure to chronic work-life stress and insufficient recovery are at high risk for developing burnout symptoms. Social services, caregiving and teaching professions with a perceived imbalance of effort and reward are often affected. Until now, a general accepted definition of burnout syndrome and its binding diagnostic criteria have not been established. Moreover, there is a strong association between chronic psychological distress and somatoform symptoms, like sleeping disturbances, headaches and abdominal pain that cannot be fully explained by medical or neurological condition. Physiologically the hypothalamus pituitary adrenal axis (HPA-axis) is the central system for the long term adaptation of an organism to stress. During stress exposure, the HPA-axis is activated and the adrenal cortex produces high levels of cortisol with a stress inhibitory function at the same time. However, exposure to long-term chronic stress is associated with biological dysregulation and can result in hypofunctioning of the HPA-axis and a state of hypocortisolism. In addition, the serotonergic system, the immune system and the amino acid metabolism get adversely affected.

Stress-related eating behaviours frequently results in an imbalance of amino acids and deficiency of micronutrients (i. e. B-vitamins and magnesium) that cause endocrine-cardiometabolic abnormalities. Intake of specific amino acids can affect the brain functioning and mental health. Some amino acids are precursors of the neurotransmitters in the brain. Moreover, l-ornithine and taurine are suggested to have an antifatigue effect. Dietary intake of B-vitamins and magnesium, the important stress-mineral, had positive effects on mood and perceived stress.

Aim of this study is to demonstrate, that the daily oral administration of a specific amino acid composition (dosage 4.2 g/day) with micronutrients (e. g. 7 vitamins of the B-complex, magnesium, zinc) designed to decrease chronic exhaustion conditions will significantly decrease the perceived chronic distress and associated chronic exhaustion conditions of women and men after 8 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Perceived Stress Questionnaire 30 (PSQ30): total score > 0.50

Exclusion Criteria:

* Age: < 18 and > 65 Years
* Perceived Stress Questionnaire (PSQ30): total score ≤ 0.50
* Supplementation or therapy with dietary supplements or drugs which contains amino acids (e. g. l-tryptophan), vitamins and other micronutrients (have to discontinue 4 weeks prior to the start of the study)
* Therapy with antidepressant drugs such as monoamine oxidase inhibitors
* Hypertension (untreated > 150/90 mmHg, treated > 140/85 mmHg)
* Organic fatigue
* Phenylketonuria
* Acute and chronic diarrhea

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Questionnaire (PSQ30) | 12-week dietary intervention
  Intervention changes in the total PSQ30 score at baseline and after 12 weeks
Perceived Stress Questionnaire (PSQ30) | 8-week dietary intervention
  Intervention changes in the total PSQ30 score at baseline and after 8 weeks

SECONDARY OUTCOMES:
Salivary cortisol concentration in the evening (between 10 and 11 pm, at least 30 minutes after dinner) and in the morning (30 minutes after waking in the morning) | 12-week dietary intervention
  Intervention changes in difference between salivary cortisol concentrations (evening - morning) at baseline and after 12 weeks
The Visual Analog Scale (VAS) | 12-week dietary intervention
  Intervention changes in mean VAS score at baseline and after 12 weeks
The Visual Analog Scale (VAS) | 8-week dietary intervention
  Intervention changes in mean VAS score at baseline and after 8 weeks

OTHER OUTCOMES:
Psychological Neurological Questionnaire (PNF) | 12-week dietary intervention
  Pre-post intervention changes in total number of points from the PNF and the psycho-neurovegetative stability (PN), a category of the PNF.
Morning salivary cortisol concentration (30 minutes after waking) | 12-week dietary intervention
  Pre-post intervention changes in salivary cortisol concentration at baseline and after 12 weeks
Evening salivary cortisol concentration (between 10 and 11 pm, at least 30 minutes after dinner) | 12-week dietary intervention
  Pre-post intervention changes in salivary cortisol concentration at baseline and after 12 weeks
3-day food records | 12-week dietary intervention
  Pre-post intervention changes in dietary intake at baseline and after 12 weeks
Endocrine-cardiometabolic parameters (i. e. serotonin, amino acids in the blood) | 12-week dietary intervention
  Pre-post intervention changes in blood parameters at baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine Metzner, Professor MD, Principal Investigator — Bonn Education Association for Dietetics r.A., Cologne, Germany
Locations (1):
- Department of Urology, University of Bonn, Bonn, Sigmund-Freud Str. 25, Germany

IPD SHARING:
Plan to Share IPD: No